CLINICAL TRIAL: NCT04758130
Title: The G.R.I.T. Study: Getting Global Rare Disease Insights Through Technology
Brief Title: Getting Global Rare Disease Insights Through Technology Study
Acronym: GRIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: M.A.G.I.C. Clinic LTD (Industry)
Collaborators: Hanalytics Solutions Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GRIT
Record Dates: First submitted 2021-01-21; First posted 2021-02-17 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Disease; Fabry Disease; Gaucher Disease; Pompe Disease; Mitochondrial Diseases
MeSH Terms: conditions — Metabolic Diseases; Fabry Disease; Gaucher Disease; Glycogen Storage Disease Type II; Mitochondrial Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Group (Experimental): Patients in this group are provided with a link to download the application and their application usage is tracked by the clinic.
  Interventions: Other: Zamplo Digital Health Platform
- Placebo Group (Placebo Comparator): Patients in this group are not provided with the clinic link to the application.
  Interventions: Other: Zamplo Digital Health Platform

INTERVENTIONS:
Other: Zamplo Digital Health Platform — This application will be provided to patients and provide them with a method to track various data related to their metabolic disease.

SUMMARY:
This project is a randomized controlled trial to use a mobile health journal, called Zamplo (formerly known as MyHealthJournal or ZoeInsights), to record patient reported outcomes (PROM) in patients with metabolic disorders.

The objective of the study is to assess the feasibility, acceptability and potential effectiveness of the Zamplo.

The primary hypothesis is as follows:

The Zamplo platform will significantly increase patient activation at 6 months post-baseline, defined as an individual's knowledge, skill, and confidence for managing their health and health care.

The primary outcome is as follows:

Patient activation following the use of Zamplo will serve as the primary outcome of interest and will be measured by the Patient Activation Measure (PAM) 13. The PAM 13 shows the degree of the patient's ability to manage their health with confidence by providing a total patient activation score.

Brief Background:

This project is a randomized controlled trial to use a mobile health journal, called Zamplo, to record patient reported outcomes (PROM) in patients with metabolic disorders.

Zamplo is a software as a service (SaaS) digital platform on both iOS and Android platforms that allows real-time entry of patient symptoms and response to medications. It provides the patients with an interface to see their progress, store questions that they will ask at the next clinic visit, record their health data and use their data to engage in their health outcomes. MAGIC Clinic Ltd., which is the largest clinic in Alberta that manages metabolic disorders such as Fabry disease, Pompe disease, and Gaucher disease, will provide access to Zamplo to patients free-of-charge to evaluate its utility in managing the symptoms of their disease.

Brief Study Design:

The study is a two-armed randomized controlled design with 1:1 allocation to treatment (Zamplo app group) or control (usual care) arms, with assessments at four time points: baseline, 1 month, 3 months (primary outcome), 6 months and 12 months follow-up post-baseline. This is an open-label trial.

The investigators intend to recruit 150 participants in this study, with 75 of them being controls.

Inclusion Criteria:

Adult patients with a diagnosis of metabolic disease Access to a smartphone with data connection Willingness to devote 10-15 mins of time in a day to log medications and notes Able to speak and write English sufficiently to complete questionnaires.

Exclusion Criteria:

Insufficient cognitive function to participate in the study The use of any electronic application requires some competency with the software on a cellphone, downloading the application and entering the data. Some patients who are elderly may not be familiar with this technology and would be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of metabolic disease
* Access to a smartphone/computer with data connection
* Willingness to devote 10-15 mins of time in a day to log medications and notes
* Able to speak and write English sufficiently to complete questionnaires

Exclusion Criteria:

* Insufficient cognitive function to participate in the study
* The use of any electronic application requires some competency with the software on a cellphone, downloading the application and entering the data. Some patients who are elderly may not be familiar with this technology and would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient Activation | 3 Months post baseline
  Patient activation following the use of Zamplo will serve as the primary outcome of interest and will be measured by the Patient Activation Measure (PAM) 13. The PAM 13 shows the degree of the patient's ability to manage their health with confidence by providing a total patient activation score. The survey will be completed by participants of the two groups at baseline and follow-up time-points.

SECONDARY OUTCOMES:
Self-Efficacy for Managing Chronic Conditions (PROMIS) | 3 Months
  Manage Medications/Treatment: Self-efficacy is defined as confidence in one's ability to successfully perform specific tasks or behaviors. Self Efficacy for Managing Chronic Conditions assesses confidence in one's ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations. Confidence in managing medication schedules of different complexity.
Patient Satisfaction | 3 Months
  This is a survey question asked during Alberta Health Quality Assessments Q11. "Thinking about all of your personal experiences within the past year with the healthcare services in Alberta that we just reviewed, to what degree are you satisfied or dissatisfied with the services you have received?"
Acceptability | 3 Months
  The acceptability of Zamplo will be assessed by patients and informal caregivers.

CONTACTS AND LOCATIONS:
Locations (1):
- M.A.G.I.C. Clinic LTD, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to request information about the study — https://magiccalgary.ca/zoeinsights/